CLINICAL TRIAL: NCT02282774
Title: Subtenon Block Combined With General Anesthesia for Vitreoretinal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Marwan Abouammoh, Associate professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-13-968
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Subtenon Anesthesia
Keywords: Vitreoretinal surgery
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB (Experimental): receive subtenon block of 4mL of 2% lidocaine and 0.5% bupivacaine (50:50) mixture
  Interventions: Drug: 2% lidocaine and 0.5% bupivacaine
- C (Sham Comparator): receive subtenon block of 4mL saline
  Interventions: Drug: Sham subtenon block

INTERVENTIONS:
Drug: 2% lidocaine and 0.5% bupivacaine — Under general anesthesia and the operating microscope, a Lieberman lid speculum was placed and the conjunctiva was cleaned with 4% povidone iodine solution. The surgeon then created a fornix-based incision through conjunctiva and tenon's tissue inferonasally midway between the insertions of the medial and inferior rectus muscles, with blunt Wescott scissors to expose the scleral surface before tunneling posteriorly with curved Stevens scissors to create a small channel to the posterior subtenon space. A blunt-tipped subtenon cannula was then inserted into the posterior subtenon space, 4mL of 2% lidocaine and 0.5% bupivacaine (50:50) mixture versus saline was introduced and the drug solution was injected slowly into the subtenon space. After administration of local anesthetic mixture, the eyelid was gently taped down, and no ocular massage was performed
  Arms: SB
Drug: Sham subtenon block
  Arms: C

SUMMARY:
To evaluate the effects of subtenon block (SB) as an adjunct to general anaesthesia on postoperative pain, oculocardiac reflex and postoperative nausea and vomiting for vitreoretinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective retinal surgery under general anesthesia

Exclusion Criteria:

* ASA physical status > Grade II,
* psychiatric conditions,
* neurological impairment,
* deafness with whom communication would be difficult in the postoperative period,
* clotting abnormalities,
* contraindications for regional anesthesia,
* drug abuse,
* history of allergy to the study drugs,
* previous vitreoretinal or strabismus surgery,
* endophthalmitis, or inflammatory eye pathology
* taking analgesics, antiemetics or drugs that might affect hemodynamics

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the time to first postoperative analgesic dose | 24 hrs
  Pain was evaluated using a VNS chart (0-no pain at all, 10-the worst pain imaginable) at 30 min, 1, 2, 4, 6, 12,18 and 24 hours postoperatively. During PACU stay, if the patient complain of pain postoperatively (VNS ≥ 4), morphine boluses of 25 µg /kg (injected at 10-min intervals) was administered intravenously if requested until the pain subsided for a maximum dose of 10 mg. At the end of 2 h, the patients were transferred from the PACU to the ward where the pain was assessed, paracetamol 15 mg/kg was given intravenously and was repeated every 4 hours if needed in the ward by a nurse who is blinded to the study group as paracetamol is the standard post-operative pain medication for patients undergoing ophthalmic surgery at our institute. Time to first post-operative analgesic, which is the time, elapsed between end of the surgical procedure and first administration of an analgesic was noted

SECONDARY OUTCOMES:
postoperative pain scores | First 24 hrs after surgery
  Pain was evaluated using a VNS chart (0-no pain at all, 10-the worst pain imaginable) at 30 min, 1, 2, 4, 6, 12,18 and 24 hours postoperatively. During PACU stay, if the patient complain of pain postoperatively (VNS ≥ 4), morphine boluses of 25 µg /kg (injected at 10-min intervals) was administered intravenously if requested until the pain subsided for a maximum dose of 10 mg. At the end of 2 h, the patients were transferred from the PACU to the ward where the pain was assessed, paracetamol 15 mg/kg was given intravenously and was repeated every 4 hours if needed in the ward by a nurse who is blinded to the study group as paracetamol is the standard post-operative pain medication for patients undergoing ophthalmic surgery at our institute. Time to first post-operative analgesic, which is the time, elapsed between end of the surgical procedure and first administration of an analgesic was noted.
number of patients requiring rescue analgesics during the 24-h study period | during the whole study (6 months)
consumption of rescue analgesics | during the whole study (6 months)
  The total number of patients receiving rescue analgesia is recorded
incidence of oculocardiac reflex | during time of surgery
incidence of postoperative nausea/vomiting | First 24 hrs after surgery
  The incidence of postoperative nausea and vomiting (PONV) was assessed by a nurse (who was blinded to the study drug) for the first 2 h in the PACU and subsequently in the ward at 6, 12 and 24 h and Only 2 possible answers was accepted (yes) or (no). Nausea was defined as subjective sensation of discomfort associated with the awareness of the urge to vomit. Vomiting was defined as a forceful expulsion of gastric contents through the mouth. Rescue antiemetic (Ondansetron 0.15 mg/kg) was given if the patient had persistent nausea or more than a single episode of vomiting or whenever patients request medication and number of patients required rescue anti-emetic postoperatively were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Abouammoh, MD, Principal Investigator — King Saud University
Locations (1):
- King Abdulaziz University Hospital at King Saud University, Riyadh, Riyadh Region, Saudi Arabia